CLINICAL TRIAL: NCT05192187
Title: Why do People With Low Back Pain Fear and Avoid Lifting?
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hasselt University (Other)
Responsible Party: Principal Investigator, Thomas Matheve, Postdoctoral researcher, Hasselt University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ThomasMatheve-2021-3
Record Dates: First submitted 2021-12-22; First posted 2022-01-14 (Actual); Last update posted 2022-02-02 (Actual); Status verified 2022-01

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain | interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- LBP (Experimental): This group will be asked to complete self-reported questionnaires on a single occasion (cross-sectional)
  Interventions: Other: Cross-sectional self-report (questionnaires)

INTERVENTIONS:
Other: Cross-sectional self-report (questionnaires) — participants in this group will be ask to complete questionnaires on one occasion (i.e., cross-sectional investigation). The questionnaires will consist of a self-developed questionnaire and standard questionnaires. The main aspects of the self-developed questionnaires are
  * perceived harmfulness of activities (selection of PHODA-SeV)
  * cognitions about lifting and pain
  * reasons for avoidance behaviour (lifting)
  Standardised questionnaires include
  * NRS for pain
  * TSK-11
  * FABQ
  * RMDQ

SUMMARY:
The investigators' main focus of this trial will be to investigate

* why people with low back pain perceive lifting (with a bent back) as harmful.
* whether general measures of pain-related fear are associated with task-specific measures of perceived harmfulness
* why people with low back pain avoid lifting (with a bent back) This will be investigated using self-report (i.e., questionnaires)

ELIGIBILITY:
Inclusion Criteria:

* low back pain >3 months

Exclusion Criteria:

* healthy persons
* low back pain <3 months

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 325 (Estimated)
Dates: Start 2022-02 (Estimated); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
cognitions about perceived harmfulness and avoidance of lifting | Day 1 (cross-sectional study)
  cognitions about perceived harmfulness and avoidance of lifting using self-developed questionnaires. Questions will be scored on a 1-5 Likert scale (1= completely disagree, 5= completely agree)

SECONDARY OUTCOMES:
Pain-related fear | Day 1 (cross-sectional study)
  Tampa Scale for Kinesiophobia 11-item version questionaire (range= 11-44. Higher score = higher levels of pain-related fear)
perceived harmfulness of specific tasks | Day 1 (cross-sectional study)
  perceived harmfulness of specific tasks measured with a selection of pictures of the Photographs of Daily Activities - Short Electronic version. Each picture will be scored on a 0-100 scale, with higher scores indicating higher levels of perceived harmfulness
Disability | Day 1 (cross-sectional study)
  Roland Morris Disability Questionnaire (score range= 0-24, higher score= higher level of disbility)
Task-specific self-efficacy | Day 1 (cross-sectional study)
  For different tasks, participants will be asked to rate the task-specific self-efficacy on a 0-10 Visual analogue scale (higher scores= higher levels of self-efficacy)
Task-specific disability | Day 1 (cross-sectional study)
  For different tasks, participants will be asked to rate their perceived disability on a 0-10 Visual analogue scale (higher scores= higher levels of disability)
Pain-related fear | Day 1 (cross-sectional study)
  Fear-Avoidance Beliefs Questionnaire. The Activity Avoidance Subscale (score range= 0-24) and Work subscale (score range= 0-42) will both be used. Higher scores indicate higher levels of pain-related fear
Pain intensity | Day 1 (cross-sectional study)
  Numeric rating scale (0-10, higher score= higher level of pain)

OTHER OUTCOMES:
Age | Day 1 (cross-sectional study)
  years
Sex | Day 1 (cross-sectional study)
  Male, female, other
Physical job requirements | Day 1 (cross-sectional study)
  Questionnaire (derived from de Dutch Musculoskeletal Questionnaire) asking about physical job requirements

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Matheve, PhD, Principal Investigator — Hasselt University
Locations (1):
- Hasselt University, Hasselt, Belgium

IPD SHARING:
Plan to Share IPD: No